CLINICAL TRIAL: NCT07241741
Title: A Single-Center Prospective Study on PTX3 as a Predictor of Insulin Resistance and Inflammatory Resolution After Bariatric Surgery
Brief Title: The Predictive Role of Preoperative Pentraxin-3 (PTX3) in Metabolic and Inflammatory Outcomes After Roux-en-Y Gastric Bypass
Acronym: PTX3-BYPASS
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Fulya Calikoglu, Lecturer, Istanbul University
Other Study IDs: ITF_2025_09
Record Dates: First submitted 2025-09-03; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Obesity; Metabolic Syndrome; Insulin Resistance; Inflammation; Roux en Y Gastric Bypass; Chronic Inflammation; C-Reactive Protein; Interleukin-6
Keywords: Pentraxin-3 (PTX3); Insulin Resistance; HOMA-IR; C-Reactive Protein (CRP); Bariatric Surgery; Roux-en-Y Gastric Bypass; Metabolic Outcomes; Inflammatory Biomarkers; Predictive Biomarker
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Insulin Resistance; Inflammation | interventions — PTX3 protein

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: High PTX3 (≥21.7 ng/mL): Participants with preoperative serum PTX3 levels ≥21.7 ng/mL. All patients underwent Roux-en-Y gastric bypass and were followed prospectively for 6 months with metabolic and inflammatory assessments.
  Interventions: Other: Biomarker Stratification by PTX3
- Group 2: Low PTX3 (<21.7 ng/mL): Participants with preoperative serum PTX3 levels <21.7 ng/mL. All patients underwent Roux-en-Y gastric bypass and were followed prospectively for 6 months with metabolic and inflammatory assessments.
  Interventions: Other: Biomarker Stratification by PTX3

INTERVENTIONS:
Other: Biomarker Stratification by PTX3 — Participants were stratified into groups according to preoperative serum PTX3 levels (≥21.7 ng/mL vs. <21.7 ng/mL). All participants underwent Roux-en-Y gastric bypass and were prospectively evaluated for metabolic (HOMA-IR, %EWL) and inflammatory (CRP, IL-6) outcomes during 6 months of follow-up.
  Other Names: Pentraxin-3 (PTX3) Grouping

SUMMARY:
This study evaluated the prognostic value of preoperative pentraxin-3 (PTX3) levels in predicting weight loss, inflammatory resolution (CRP, IL-6), and metabolic improvements (HOMA-IR) following Roux-en-Y gastric bypass in patients with obesity.

DETAILED DESCRIPTION:
This single-center longitudinal study was conducted at Istanbul University Hospital. A total of 23 patients undergoing primary Roux-en-Y gastric bypass were included. PTX3 levels were measured preoperatively, and patients were stratified according to a data-derived cut-off (~21.7 ng/mL). Outcomes assessed at baseline, 3 months, and 6 months included body weight, BMI, excess weight loss (%EWL), fasting insulin, HOMA-IR, CRP, and IL-6. The primary hypothesis was that preoperative PTX3 would predict postoperative CRP normalization and insulin resistance improvement.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years
* Body mass index (BMI) ≥40 kg/m², or BMI ≥35 kg/m² with obesity-related comorbidity
* Eligible for primary Roux-en-Y gastric bypass
* Able to provide written informed consent

Exclusion Criteria:

* Previous bariatric surgery
* Severe hepatic, renal, or cardiac failure
* Active infection or inflammatory disease
* Malignancy

Ages: 18 Days to 65 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Adults with obesity scheduled to undergo primary Roux-en-Y gastric bypass at Istanbul University Hospital.
  Sexes Eligible for Study: All Gender-Based: No Accepts Healthy Volunteers: No
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Change in HOMA-IR from baseline to 6 months | Baseline, 3 months, 6 months
  Assessment of the improvement in insulin resistance after Roux-en-Y gastric bypass, measured by the homeostasis model assessment of insulin resistance (HOMA-IR). Preoperative PTX3 stratification will be used to evaluate predictive value.

SECONDARY OUTCOMES:
Percent Excess Weight Loss (%EWL) at 6 months | 6 months
  Evaluation of weight loss outcomes after surgery, calculated as percent excess weight loss (%EWL). Comparisons will be made between PTX3 high vs. low groups.
CRP normalization at 6 months | 6 months
  Proportion of patients achieving CRP ≤5 mg/L after surgery. Predictive value of baseline PTX3 will be assessed.
Change in IL-6 from baseline to 6 months | Baseline, 3 months, 6 months
  Change in serum IL-6 levels after surgery, analyzed between PTX3 high vs. low groups.

IPD SHARING:
Plan to Share IPD: No
The study team does not plan to share individual participant data at this time.